CLINICAL TRIAL: NCT01908023
Title: Exercise and Radiotherapy, a Good Combination? A Pilot Study of Group Exercise for Patients With Breast Cancer
Brief Title: Exercise and Radiotherapy, a Good Combination?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/271
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Breast Neoplasms
Keywords: exercise therapy; oxygen consumption
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise (Experimental)
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — One hour, twice a week, for 5 weeks: warming-up with aerobic exercises, endurance exercises, strength exercises for large muscle groups, body awareness, range-of- motion exercises for the shoulders and stretching and relaxation

SUMMARY:
Every year, almost 3000 Norwegian women are diagnosed with breast cancer. Various symptoms of short-and long-term side effects may be experienced, such as physical deterioration, reduced quality of life and fatigue. At St.Olavs Hospital, Trondheim University Hospital, all out-patients undergoing post operative radiotherapy are currently offered participation in group exercise training sessions. The main purpose of this study is to evaluate these out-patient group exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

* Surgery for breast cancer.
* Completed chemotherapy treatment.
* Radiotherapy is scheduled.

Exclusion Criteria:

* metastatic disease
* pregnancy
* drug abuse

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
changes in physical performance | from baseline to 6 weeks
  aerobic capacity (VO2peak)

SECONDARY OUTCOMES:
perceived coping | from baseline to 6 weeks
  Patient Activation Measure (PAM)
Range of motion | from baseline to 6 weeks
quality of life | from baseline to 6 weeks
  questionnaire SF-36
activity level | from baseline to 6 weeks
  International physical activity questionnaire
balance | from baseline to 6 weeks
  Functional Reach

CONTACTS AND LOCATIONS:
Overall Officials: Inger L Aamot, phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Klinikk for Kliniske Servicefunksjoner, Trondheim, Norway